CLINICAL TRIAL: NCT01620775
Title: MR (Magnetic Resonance) Imaging of the Excitatory and Inhibitory Neurotransmitters in Chronic Pain
Brief Title: MR(Magnetic Resonance) Imaging of Neurotransmitters in Chronic Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator was unable to fulfill his responsibilities.
Sponsor: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00055261
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Chronic Low Back Pain; Diabetic Peripheral Neuropathy; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (4):
- Knee osteoarthritis (MRI, surveys, pain testing) (Experimental): Subjects previously diagnosed with knee osteoarthritis will have an MRI with imaging that measures brain metabolites. There are surveys to complete and a session of pain tolerance testing.
  Interventions: Other: MRIs; Other: Pain testing
- Healthy controls (MRI, surveys,pain testing) (Active Comparator): Healthy volunteers will have an MRI with imaging that measures brain metabolites. There are surveys to complete and a session of pain tolerance testing.
  Interventions: Other: MRIs; Other: Pain testing
- diabetic peripheral neuropathy (Experimental): Subjects previously diagnosed with diabetic peripheral neuropathy will have an MRI with imaging that measures brain metabolites. There are surveys to complete and a session of pain tolerance testing.
  Interventions: Other: MRIs; Other: Pain testing
- chronic low back pain (Experimental): Subjects previously diagnosed with chronic low back pain will have an MRI with imaging that measures brain metabolites. There are surveys to complete and a session of pain tolerance testing.
  Interventions: Other: MRIs; Other: Pain testing

INTERVENTIONS:
Other: MRIs — Subjects will have an MRI scan to view specific images, and brain activity patterns thought to be affected in patients with KOA, chronic low back pain and diabetic patients with painful neuropathy. Healthy volunteers will undergo the same MRI scan that lasts about 90 min.
Other: Pain testing — There will be a 1-1.5 hour session including pain tolerance testing.

SUMMARY:
This study is designed to assess:

Hypothesis #1: That there is a significant central pain component in a distinct subset of patients diagnosed with knee osteoarthritis(KOA), Chronic low back pain(CLBP), painful diabetic neuropathy(PDN.)

Hypothesis # 2: To establish a reliable strategy for differentiation of central pain predominant from peripheral pain predominant knee osteoarthritis(KOA), chronic low back pain(CLBP)and peripheral diabetic neuropathy(PDN) patients using clinical features, experimental pain testing and magnetic resonance(MR) Spectroscopy.

DETAILED DESCRIPTION:
This study will identify clinical and neuroimaging markers in chronic pain in an effort to provide individual-based treatments. This study will differentiate chronic pain subjects (knee osteoarthritis, low back pain and painful diabetic neuropathy) into two groups: those who have central pain predominant symptoms and those who have peripheral pain predominant symptoms. The response to medical treatment between these two groups is quite different, thus a reliable strategy to correctly categorize chronic pain sufferers offers the opportunity to provide targeted, effective treatments. Chronic pain is a prevalent problem in the VA veteran population with significant associated costs; in particular knee osteoarthritis, chronic low back pain and painful diabetic neuropathy are common in this population. The proposed study will use different clinical pain tests and advanced neuroimaging techniques to improve our understanding of chronic pain and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Must be Right Handed.

(Chronic Pain with knee osteoarthritis)

* Diagnosed with: unilateral, symptomatic knee osteoarthritis based on American College of Rheumatology (ACR) criteria.
* Have had a knee x-ray within the last 6 months.
* Must have average pain intensity of 4 or greater on a 0 (no pain) to 10 (worst pain imaginable) scale.

(Chronic Low Back Pain)

* Have primary complaint of constant or intermittent back pain of at least 6 months duration.
* Have a Roland Morris Disability Questionnaire score of >7.

(Diabetes Mellitus with Painful Peripheral Neuropathy)

* Have a diagnosis of diabetes mellitus for at least 6 months.
* Have a diagnosis of diabetic peripheral neuropathy.
* Have had Electromyography(EMG) testing within the last 6 months.
* Have a >40 mm score on the short-form McGill Pain questionnaire.

(Healthy controls)

* Must be pain free
* No history of neurological or psychiatric illness.
* No diagnosis of Diabetes Mellitus.
* No evidence of neuropathy on clinical assessment.

Exclusion Criteria:

* Being pregnant.
* Have metal in the body or other contraindications to Magnetic Resonance Imaging (MRI).
* Have a chronic pain condition unrelated to knee osteoarthritis, chronic low back pain or diabetes.
* Have currently or a history of brain infection, stroke or tumor.
* Have a risk factor for other non-diabetic neuropathies

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-09; Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

PRIMARY OUTCOMES:
Assessment of chronic pain | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Foerster Bradley, M.D., Principal Investigator — University of Michigan; Bradley Foerster, M.D., Principal Investigator — University of Michigan
Locations (1):
- VA Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No